CLINICAL TRIAL: NCT03603340
Title: Efficacy, Safety and Toxicology of Electronic Nicotine Delivery Systems as an Aid for Smoking Cessation (ESTxENDS Trial)- the Depression Substudy of ESTxENDS
Brief Title: The ESTxENDS Trial- Substudy on the Effects of Using Electronic Nicotine Delivery Systems (ENDS) on Depression
Acronym: ESTxENDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Lausanne (Other); University of Geneva, Switzerland (Other); University of Zurich (Other); State Hospital, St. Gallen (Other Government); Swiss National Science Foundation (Other); Krebsforschung Schweiz, Bern, Switzerland (Other); Federal Office of Public Health, Switzerland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-02332f
Record Dates: First submitted 2018-07-02; First posted 2018-07-27 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation; Depression
MeSH Terms: conditions — Smoking Cessation; Depression

STUDY DESIGN:
Masking Description: Statisticians and laboratory personnel will be blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: ENDS (vaporizer/e-cig) and smoking cessation counseling
- Control group (Active Comparator)
  Interventions: Other: Smoking cessation counseling

INTERVENTIONS:
Other: ENDS (vaporizer/e-cig) and smoking cessation counseling — Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Intervention group
Other: Smoking cessation counseling — Participants in the control group will receive smoking cessation counseling only. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Control group

SUMMARY:
--> This is a substudy of the main ESTxENDS trial (NCT03589989). Depression outcomes should be considered secondary outcomes of the main smoking cessation outcome formulated in NCT03589989.

Cigarette smoking is the leading cause of preventable death in Switzerland and still more than a quarter of the Swiss population smokes cigarettes. Smoking and depression are strongly associated. Individuals with depression are twice as likely to be smokers than persons without a depression. Studies have shown that attempts to quit tobacco smoking are more likely to fail for individuals with depression than without. Depressive symptoms are common in prolonged nicotine withdrawal and individuals with depression are more nicotine dependent and more likely to suffer depressive symptoms during nicotine withdrawal compared to smokers in the general population.

Recently, electronic nicotine delivery systems (ENDS; also called vaporizer or electronic cigarette) have become popular with smokers who want to stop smoking or reduce their exposure to inhaled chemicals since ENDS use appears to be safer than tobacco smoking. ENDS with nicotine containing e-liquids may be effective in assisting with tobacco smoking cessation without suffering depressive symptoms.

This study will therefore test the efficacy of ENDS for cigarette smoking cessation, the safety of ENDS on adverse events and the effect of ENDS on health-related outcomes such as depression and exposure to inhaled chemicals.

For the main ESTxENDS trial (NCT03589989), cigarette smokers motivated to quit smoking cigarettes will be included. Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants in the control group will receive smoking cessation counseling only. All participants will be followed over a 24-month period. Presence and severity of depression will be assessed using the 9-question depression scale from the patient health questionnaire (PHQ-9) at baseline and at 6, 12 and 24 months' follow-up.

ELIGIBILITY:
Inclusion criteria:

* Informed Consent as documented by signature
* Persons aged 18 or older
* Currently smoking 5 or more cigarettes a day for at least 12 months
* Willing to try to quit smoking within the next 3 months,
* Persons providing a valid phone number, a valid email address and/or a valid postal address.

Exclusion criteria:

* Known hypersensitivity or allergy to contents of the e-liquid
* Participation in another study with investigational drug within the 30 days preceding the baseline visit and during the present study where interactions are to be expected
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the scheduled study intervention, i.e. within the first 6-months of the study
* Persons having used ENDS or tobacco heating systems regularly in the 3 months preceding the baseline visit
* Persons having used nicotine replacement therapy (NRT) or other medications with demonstrated efficacy as an aid for smoking cessation such as varenicline or bupropion within the 3 months preceding the baseline visit
* Persons who cannot attend the 6- month follow-up visit for any reason
* Cannot understand instructions delivered in person or by phone, or otherwise unable to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Assessment of severity of self-reported symptoms of depression_1 | 6 months post quit date
  Measured using the 9-question depression scale from the patient health questionnaire (PHQ-9). The PHQ-9 is it is used to monitor the severity of depression. The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
Assessment of severity of self-reported symptoms of depression_2 | 12 months post quit date
  Measured using the 9-question depression scale from the patient health questionnaire (PHQ-9). The PHQ-9 is it is used to monitor the severity of depression. The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
Assessment of severity of self-reported symptoms of depression_3 | 24 months post quit date
  Measured using the 9-question depression scale from the patient health questionnaire (PHQ-9). The PHQ-9 is it is used to monitor the severity of depression. The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).

SECONDARY OUTCOMES:
Assessment of change of severity of self-reported symptoms of depression | Change from baseline to 6,12, 24 months post quit date
  Measured using the 9-question depression scale from the patient health questionnaire (PHQ-9). The PHQ-9 is it is used to monitor the severity of depression. The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).

CONTACTS AND LOCATIONS:
Overall Officials: Reto Auer, Prof.Dr.med, Study Director — Berner Institut für Hausarztmedizin (BIHAM)
Locations (5):
- Switzerland (5):
  - Unisanté, Centre universitaire de médecine générale et santé publique, Université de Lausanne, Lausanne, Canton of Vaud
  - University Clinic for General Internal Medicine, Bern University Hospital, Bern
  - Département de médecine interne, Hôpitaux universitaires de Genève, Geneva
  - Lungenzentrum, Klinik für Pneumologie und Schlafmedizin, Kantonsspital St. Gallen, Sankt Gallen
  - Epidemiology, Biostatistics and Prevention Institute (EBPI), University of Zurich, Zurich

REFERENCES:
- [Background] Hall SM, Humfleet GL, Munoz RF, Reus VI, Robbins JA, Prochaska JJ. Extended treatment of older cigarette smokers. Addiction. 2009 Jun;104(6):1043-52. doi: 10.1111/j.1360-0443.2009.02548.x. Epub 2009 Apr 9. PMID 19392908
- [Background] Kalman D, Morissette SB, George TP. Co-morbidity of smoking in patients with psychiatric and substance use disorders. Am J Addict. 2005 Mar-Apr;14(2):106-23. doi: 10.1080/10550490590924728. PMID 16019961
- [Background] Lasser K, Boyd JW, Woolhandler S, Himmelstein DU, McCormick D, Bor DH. Smoking and mental illness: A population-based prevalence study. JAMA. 2000 Nov 22-29;284(20):2606-10. doi: 10.1001/jama.284.20.2606. PMID 11086367
- [Background] Ziedonis D, Hitsman B, Beckham JC, Zvolensky M, Adler LE, Audrain-McGovern J, Breslau N, Brown RA, George TP, Williams J, Calhoun PS, Riley WT. Tobacco use and cessation in psychiatric disorders: National Institute of Mental Health report. Nicotine Tob Res. 2008 Dec;10(12):1691-715. doi: 10.1080/14622200802443569. PMID 19023823
- [Background] Glassman AH. Cigarette smoking: implications for psychiatric illness. Am J Psychiatry. 1993 Apr;150(4):546-53. doi: 10.1176/ajp.150.4.546. PMID 8465868
- [Background] Weinberger AH, Pilver CE, Desai RA, Mazure CM, McKee SA. The relationship of major depressive disorder and gender to changes in smoking for current and former smokers: longitudinal evaluation in the US population. Addiction. 2012 Oct;107(10):1847-56. doi: 10.1111/j.1360-0443.2012.03889.x. Epub 2012 May 17. PMID 22429388
- [Background] Bolam B, West R, Gunnell D. Does smoking cessation cause depression and anxiety? Findings from the ATTEMPT cohort. Nicotine Tob Res. 2011 Mar;13(3):209-14. doi: 10.1093/ntr/ntq244. Epub 2011 Feb 17. PMID 21330275
- [Background] Gierisch JM, Bastian LA, Calhoun PS, McDuffie JR, Williams JW Jr. Smoking cessation interventions for patients with depression: a systematic review and meta-analysis. J Gen Intern Med. 2012 Mar;27(3):351-60. doi: 10.1007/s11606-011-1915-2. Epub 2011 Oct 26. PMID 22038468
- [Background] Weinberger AH, Mazure CM, Morlett A, McKee SA. Two decades of smoking cessation treatment research on smokers with depression: 1990-2010. Nicotine Tob Res. 2013 Jun;15(6):1014-31. doi: 10.1093/ntr/nts213. Epub 2012 Oct 25. PMID 23100459
- [Derived] Rihs A, Schoeni A, Scharf T, Jakob J, Tal K, Jacot-Sadowski I, Humair JP, Frei A, Brutsche M, Rodondi N, Auer R, Baggio S. Effect of e-cigarettes for smoking cessation on depressive and anxiety symptoms: Secondary analysis of a randomized controlled trial. Gen Hosp Psychiatry. 2025 Mar-Apr;93:67-72. doi: 10.1016/j.genhosppsych.2025.01.011. Epub 2025 Jan 16. PMID 39827790